CLINICAL TRIAL: NCT05803954
Title: Mulligan Mobilization Technique Versus Neural Mobilization on Nerve Root Function in Patients With Cervical Radiculopathy: Randomized Controlled Trial
Brief Title: Mobilization With Movement vs. Neural Mobilization on Nerve Root Function in Patients With Cervical Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amany Ismail Elmetwaly Selem, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMNM2023
Record Dates: First submitted 2023-03-25; First posted 2023-04-07 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Disc Herniation; Cervical Radiculopathy; Cervical Radiculopathy at C5 Nerve Root; Cervical Radiculopathy at C6 Nerve Root; Cervical Radiculopathy at C7 Nerve Root
MeSH Terms: conditions — Intervertebral Disc Displacement; Radiculopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (SNAGs group) (Experimental)
  Interventions: Other: Sustained natural apophyseal glides (SNAGS); Other: Traditional physical therapy
- Group B (Neural mobilization group) (Experimental)
  Interventions: Other: Neural mobilization; Other: Traditional physical therapy
- Group C (traditional physical therapy) (Active Comparator)
  Interventions: Other: Traditional physical therapy

INTERVENTIONS:
Other: Sustained natural apophyseal glides (SNAGS) — SNAGS will be applied with the patient sitting comfortably on a stool. The therapist stand behind the patient and the medial border of one thumb's distal phalanx is placed on the articular pillar on the chosen side of the suspected site of lesion. The thumb nail slope at approximately 45 degree (in the direction of the eyeball). SNAGS mulligan will be given by active movement followed by passive overpressure based on the movement restricted by frequency of treatment will be three sets of ten repetitions. SNAG the anteroposterior mobilization of the second cervical vertebrae is sustained for 10 to 30 s depending on response. A maximum of 6 repetitions will be given if there is a reduction in headache intensity at the time of the first application. A total of 20 oscillations (1 oscillation/1 second) will be given to each joint with a total duration of 15 minutes
  Arms: Group A (SNAGs group)
Other: Neural mobilization — Neural mobilization will be applied with grade three neural mobilization and traditional therapy: Subjects will be placed in supine position and remained relaxed with the feet uncrossed. The patient will be slightly angled obliquely for easier access to the scapula. The therapist will be depressed the scapula with concomitant upper extremity joint positioning as per median nerve bias i.e., ULTT2 (shoulder abduction, elbow extension with forearm supination, wrist and fingers extended and ulnar deviated and thumb abduction). The wrist will be used as a tension factor and at the point where tension was felt by the therapist and perceived by the subject. Grade 3 oscillations were given rhythmically and slowly to each joint from proximal to distal. A total of 20 oscillations (1 oscillation/1 second) were given to each joint with a total duration of 15 minutes.
  Arms: Group B (Neural mobilization group)
Other: Traditional physical therapy — traditional therapy will be applied in the form of stretching for bilateral upper and middle trapezius muscles and bilateral neck rotators and isometric strengthening exercises for neck rotators, extensors, side bending muscles. Exercise was repeated for ten repetitions per session. In addition to hot pack was placed over the neck and upper part of shoulders musculature. This was being applied for ten min, over middle trapezius trigger Point itself.

SUMMARY:
This study will be conducted to compare the effect of sustained natural apophyseal glides (SNAGS) versus neural mobilization on clinical outcomes such as 1- nerve root function in the form of: (A) peak to peak amplitude; (B) latency; (C) F wave. 2- pain pressure threshold (PPT) and 3- Neck disability index (NDI) in patients with cervical disc (C5-C6 and/or C6-C7) herniation.

Seventy two patients from both gender with cervical disc (C 5-C 6 and/or C 6- C7) herniation with both sensory and motor nerve affections will be recruited for this study following referral from an experienced neurologist and confirmed diagnosis by MRI. The patients' age will range between 20-50 years, body mass index (BMI) from 18 to 25 kg/cm2.

The patients will be assigned randomly by permuted block to three equal groups; group (A) will receive SNAGS in addition to traditional therapy, group (B) will receive neural mobilization in addition to traditional therapy and group (C) will receive traditional therapy.

peak to peak amplitude, nerve latency and F wave will be measured by electromyography, , pressure pain threshold will be measured by commander algometer. Neck disability will be measured by Arabic neck disability index.

ELIGIBILITY:
Inclusion Criteria:

1. seventy patients with cervical disc (C 5-C 6 and/or C 6- C7) herniation with both sensory and motor nerve affections, referred from neurologist and confirmed diagnosis by MRI
2. Both sexes.
3. Age between 20-50 years.
4. Patients with neck pain radiating down to the arm.
5. Patients with positive findings for spurling test, Upper Limb Tension Test One (ULTTO), cervical distraction test and cervical rotation test towards the symptomatic side <60.
6. BMI from 18 to 25 kg/cm2
7. Existed active trigger points within middle trapezius and/ or cervical region.
8. Positive Pittsburgh sleep quality index' value >10, means moderate and/ or sever difficulty.

Exclusion Criteria:

1. Patients experiencing primary shoulder or upper extremity problem of local origin
2. cardiovascular disorders and respiratory disorders,
3. pathological conditions involving cervical spine like vertebro basilar insufficiency and canal stenosis
4. osteophytes in cervical vertebrae
5. Patients who were undergoing treatment for neck pain with other means of physiotherapy at the time of the study
6. Cervical fractures, spinal surgery or other spinal pathologies (i.e. ankylosing spondylitis, spondylolisthesis)
7. Peripheral nerve lesions like neurotmesis and axonotmesis.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
F-wave parameters | Change over the course of the study, from baseline to the end of treatment program at 4 weeks
  Evaluation of the spinal motoneuron excitability through the measurement of the F wave parameters
Somatosensory Evoked Potentials (SEPs) Latency and Amplitude | Change over the course of the study, from baseline to the end of treatment program at 4 weeks
  SEPs are the electrical signals generated by the nervous system in response to somatosensory stimuli. SEPs are read on the skull with electroencephalography (EEG)
Pain pressure threshold by Pressure algometer | Change over the course of the study, from baseline to the end of treatment program at 4 weeks
  An algometer will be used used to quantify pain intensity by pressure

SECONDARY OUTCOMES:
Neck disability Index | Change over the course of the study, from baseline to the end of treatment program at 4 weeks
  Methods of assessment for such disability, especially those targeted at activities of daily living which are most affected by neck pain, questionnaire 10-item scaled entitled the Neck Disability Index (NDI)

CONTACTS AND LOCATIONS:
Overall Officials: Amany I. Selem, BSc, Principal Investigator — Cairo University
Locations (1):
- Ismailia medical complex, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No